CLINICAL TRIAL: NCT05488028
Title: Three-dimensional Facial Swelling Evaluation of Piezo-electric Versus Conventional Drilling Bur Surgery of Impacted Lower Third Molar: a Randomized Clinical Trial
Brief Title: 3D Evaluation of Facial Swelling Post Impacted Lower Third Molars Surgery: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01-20
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Swelling/ Edema; Impacted Third Molar Tooth
Keywords: piezosurgery; conventional osteotomy; impacted lower third molar; facial scan; 3d rendering
MeSH Terms: conditions — Edema

STUDY DESIGN:
Intervention Model Description: Split-mouth model
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezosurgery (Experimental): Patients needing lower third molar surgery, in which the osteotomy is performed by the use of a piezo-electric instrument
  Interventions: Procedure: Piezo-electric surgery of impacted lower third molars
- Conventional bur (Experimental): Patients needing lower third molar surgery, in which the osteotomy is performed by the use of a drilling bur
  Interventions: Procedure: Rotary bur surgery of impacted lower third molars

INTERVENTIONS:
Procedure: Piezo-electric surgery of impacted lower third molars — During lower third molar surgery, osteotomy is performed using piezoelectric instrumentation.
  When necessary, tooth sectioning was performed with a high-speed tungsten carbide slit drill under saline irrigation and the tooth removed in single or multiple segments.
  Arms: Piezosurgery
Procedure: Rotary bur surgery of impacted lower third molars — During lower third molar surgery, osteotomy is performed using rotary instruments
  Arms: Conventional bur

SUMMARY:
Aim of the study is to evaluate the swelling following the osteotomy when performed with drilling bur versus piezo-electric instrument in the mandibular impacted third molar extraction, using a facial reconstruction software

ELIGIBILITY:
Inclusion Criteria:

* good general health conditions;
* presence of bilateral and symmetrical impacted third molars (according to the classifications of Winter and Pell and Gregory);

Exclusion Criteria:

* no clinical evidence of major facial asymmetry;
* use of medication that would influence or alter wound healing;
* temporomandibular joint disorder history;
* smoking

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Facial swelling | 7 days
  T0-T1 and T0-T2 scans are opened and superimposed through three reference points:
  endocanthion left (inner most point on commissure of left eye fissure), endocanthion right (inner most point on commissure of right eye fissure) and subnasale (mid point of columella).
  After matching, the swelling was calculated by selecting the area of the swelling and subtracting the two images.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Policlinic Gaetano Martino, Messina, Messina (ME), Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caputo A, Rubino E, Marciano A, Peditto M, Bellocchio AM, Nucera R, Oteri G. Three-dimensional facial swelling evaluation of piezo-electric vs conventional drilling bur surgery of impacted lower third molar: a randomized clinical trial. BMC Oral Health. 2023 Apr 21;23(1):233. doi: 10.1186/s12903-023-02910-6. PMID 37085833